CLINICAL TRIAL: NCT06551350
Title: Retrospective Assessment of Referral of a Major Trauma Patient in Val-d'Oise
Brief Title: Retrospective Assessment of Referral of a Major Trauma Patient
Acronym: SAMU-TRAUMAS
Status: Recruiting | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0924
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Trauma Injury
Keywords: Major trauma; Mobile Intensive Care Unit (MCIU)
MeSH Terms: conditions — Accidental Injuries | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data Collection — Collection of medical data from MICU intervention file and the medical records of patients at the destination hospital

SUMMARY:
The aim of this study is to find out whether major trauma patients from the Val d'Oise are referred to the appropriate trauma centre for their care and to assess the quality of triage within the Val d'Oise department.

DETAILED DESCRIPTION:
In France, the number of major trauma is estimated at between 15,000 and 20,000 per year. It is the leading cause of death in patients under the age of 40, and is a significant source of long-term dependency. Mortality from severe trauma varies depending on the region and the circumstances of the accident. Effective initial care and referral to specialist trauma centres are crucial to improving survival. Access to these centres must be guaranteed throughout France. Trauma centres play a central role in the management of serious trauma patients. They are classified by level, from level I to level III.

The triage process aims to direct the patient to the trauma centre with the appropriate level of care. The challenge is to send the "right patient to the right place at the right time". Over-triage and under-triage are two critical concepts in the management of trauma patients. Over-triage (patients considered to be more seriously injured than they really are) leads to excessive consumption of resources and increases waiting times for patients who really need a level I or II trauma centre. Under-triage (patients considered to be less seriously injured than they really are), is characterised by patients being referred to a trauma centre that is insufficiently equipped for their needs, compromises their chances of survival and recovery. In both cases, the loss of chance for the patient is real.

The aim of this study is to find out whether major trauma patients from the Val d'Oise are referred to the appropriate trauma centre for their care, and to assess the quality of triage within the Val d'Oise department.

ELIGIBILITY:
Inclusion Criteria :

* Between the 1st January 2023 and the 31th December 2023
* Regulated by SAMU 95 with suspected major trauma
* Sending an MCIU
* At least 1 Vittel criterion*

Exclusion Criteria :

* Death on site
* Care by an MICU team outside the 95
* Minor patients and legal protection
* Transport refusals

  * Vittel criterion :

    • Physiological variables : Glasgow score < 13 Systolic blood pressure < 90 mmHg O2 saturation < 90%

    • Elements of kinetics : Ejection from a vehicle Other passenger killed in the same vehicle Fall > 6 metres Victim thrown or crushed Overall assessment (deformation of the vehicle, estimated speed, absence of helmet, absence of seatbelt) Blast

    • Anatomical lesions : Penetrating trauma to the head, neck, thorax, abdomen, pelvis, arm or thigh Flail chest Severe burn, smoke inhalation Pelvic fracture Suspected spinal cord injury Amputation of wrist, ankle or above Acute limb ischaemia

    • Pre-hospital resuscitation : Assisted ventilation Filling > 1000 ml with colloids Catecholamines Inflated shock-proof trousers

    • Medical context (to be assessed) : Age > 65 Cardiac or coronary insufficiency Respiratory insufficiency Pregnancy (2nd and 3rd trimesters) Blood crase disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients regulated by SAMU 95 with suspected major trauma between the 1st January 2023 and the 31th December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 461 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Triage assessment of a major trauma patient | At the end of the study, an average of 9 month
  The criterion is the evaluation of the referral of the major trauma patient after post-Medics injury assessment into over, normo and under-triage
  The over-triage patient is referred to a level I trauma centre with an Injury Severity Score (ISS) <16
  The normo-triage patients are either referred to:
  * a level 1 trauma centre with an ISS >15
  * the local scanner and then to an intensive care unit at the scanner site
  * in the emergency department and then to a surgical unit
  * emergency with a return home afterwards
  The under-triage patient is either referred to:
  * the local scanner and then to a level 1 trauma centre
  * initially emergency with hospitalisation in an intensive care or continuing care unit afterwards

SECONDARY OUTCOMES:
Assess if the intervention time is correlated with an under-triage | At the end of the study, an average of 9 month
  The correlation will be assessed by the proportion of patients under-triaged during the following hours:
  * 7am to 9am
  * From 6pm to 9pm
  * From 9pm to 7am i.e. the ratio between the number of under-triaged patients and the number of major trauma patients treated during the defined time slots.
Assess if presumed alcohol intoxication is correlated with a higher rate of under-triage | At the end of the study, an average of 9 month
  The correlation will be assessed by the proportion of patients under-triaged in patients with suspected alcohol intoxication. Presence of suspected alcohol intoxication assessed clinically i.e. the ratio between the number of under-triaged patients with suspected alcohol intoxication and the total number of major trauma patients
Assess if deliberate toxic poisoning is correlated with a higher rate of under-triage | At the end of the study, an average of 9 month
  The correlation will be assessed by the proportion of patients under-triaged in patients with suspected deliberate toxic poisoning. Presence of deliberate toxic poisoning assessed clinically i.e. the ratio between the number of under-triaged patients with suspected deliberate toxic poisoning and the total number of major trauma patients
Assess if the TRENAU grade is predictive in pre-hospital of an appropriate referral following an intra-hospital trauma assessment | At the end of the study, an average of 9 month
  The criterion will be assessed by the correlation between TRENAU grade and level of trauma centre for final admission :
  TRENAU A in a level 1 trauma centre TRENAU B in a level 2 trauma centre TRENAU C in a level 3 trauma centre The TRENAU grade (Trauma System du Réseau Nord Alpin des Urgences) is used to classify major trauma patients into 3 categories (A, B and C) in the pre-hospital phase, so that they can be referred to the appropriate level of hospital
Assess if the positive Shock-Index is predictive of an appropriate pre-hospital referral to a level 1 trauma centre | At the end of the study, an average of 9 month
  The criterion will be assessed by the number of patient with positive Shock-Index (≥ 0.9) at the time of MCIU care referred to a level 1 trauma centre (final admission)
Assess if the positive Shock-Index ( ≥ 0.9 ) is predictive of an intra-hospital blood transfusion | At the end of the study, an average of 9 month
  The criterion will be assessed by the number of patient with positive Shock-Index (≥ 0.9) at the time of MCIU care and who have had an intra-hospital blood transfusion
Assess if the MGAP is predictive of an appropriate referral following an intra-hospital trauma assessment | At the end of the study, an average of 9 month
  The evaluation criterion will be assessed as follow :
  Number of patient with a MGAP between 23 and 29 and an final admission in a level 3 trauma centre Number of patient with a MGAP between 18 and 22 and an final admission in a level 2 trauma centre Number of patient with a MGAP < 18 and an final admission in a level 3 trauma centre The MGAP score (Mechansim, Glasgow, Age, Arterial pressure) can predict the risk of in-hospital death in trauma patients. Three risk groups have been defined: low (23-29 points), intermediate (18-22 points) and high (<18 points).

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice LOUVET, Principal Investigator — Hôpital NOVO
Locations (1):
- Resuscitation Services (SAMU 95/SMUR) - Hôpital NOVO -Pontoise Site, Pontoise, France

REFERENCES:
- [Background] MacKenzie EJ, Rivara FP, Jurkovich GJ, Nathens AB, Frey KP, Egleston BL, Salkever DS, Scharfstein DO. A national evaluation of the effect of trauma-center care on mortality. N Engl J Med. 2006 Jan 26;354(4):366-78. doi: 10.1056/NEJMsa052049. PMID 16436768
- [Background] Haagsma JA, Graetz N, Bolliger I, Naghavi M, Higashi H, Mullany EC, Abera SF, Abraham JP, Adofo K, Alsharif U, Ameh EA, Ammar W, Antonio CA, Barrero LH, Bekele T, Bose D, Brazinova A, Catala-Lopez F, Dandona L, Dandona R, Dargan PI, De Leo D, Degenhardt L, Derrett S, Dharmaratne SD, Driscoll TR, Duan L, Petrovich Ermakov S, Farzadfar F, Feigin VL, Franklin RC, Gabbe B, Gosselin RA, Hafezi-Nejad N, Hamadeh RR, Hijar M, Hu G, Jayaraman SP, Jiang G, Khader YS, Khan EA, Krishnaswami S, Kulkarni C, Lecky FE, Leung R, Lunevicius R, Lyons RA, Majdan M, Mason-Jones AJ, Matzopoulos R, Meaney PA, Mekonnen W, Miller TR, Mock CN, Norman RE, Orozco R, Polinder S, Pourmalek F, Rahimi-Movaghar V, Refaat A, Rojas-Rueda D, Roy N, Schwebel DC, Shaheen A, Shahraz S, Skirbekk V, Soreide K, Soshnikov S, Stein DJ, Sykes BL, Tabb KM, Temesgen AM, Tenkorang EY, Theadom AM, Tran BX, Vasankari TJ, Vavilala MS, Vlassov VV, Woldeyohannes SM, Yip P, Yonemoto N, Younis MZ, Yu C, Murray CJ, Vos T. The global burden of injury: incidence, mortality, disability-adjusted life years and time trends from the Global Burden of Disease study 2013. Inj Prev. 2016 Feb;22(1):3-18. doi: 10.1136/injuryprev-2015-041616. Epub 2015 Dec 3. PMID 26635210
- [Background] Hirsch M, Carli P, Nizard R, Riou B, Baroudjian B, Baubet T, Chhor V, Chollet-Xemard C, Dantchev N, Fleury N, Fontaine JP, Yordanov Y, Raphael M, Burtz CP, Lafont A; health professionals of Assistance Publique-Hopitaux de Paris (APHP). The medical response to multisite terrorist attacks in Paris. Lancet. 2015 Dec 19;386(10012):2535-8. doi: 10.1016/S0140-6736(15)01063-6. Epub 2015 Nov 28. No abstract available. PMID 26628327
- [Background] Cotte J, Courjon F, Beaume S, Prunet B, Bordes J, N'Guyen C, Contargyris C, Lacroix G, Montcriol A, Kaiser E, Meaudre E. Vittel criteria for severe trauma triage: Characteristics of over-triage. Anaesth Crit Care Pain Med. 2016 Apr;35(2):87-92. doi: 10.1016/j.accpm.2015.06.013. Epub 2015 Dec 1. PMID 26592159
- [Background] Sartorius D, Le Manach Y, David JS, Rancurel E, Smail N, Thicoipe M, Wiel E, Ricard-Hibon A, Berthier F, Gueugniaud PY, Riou B. Mechanism, glasgow coma scale, age, and arterial pressure (MGAP): a new simple prehospital triage score to predict mortality in trauma patients. Crit Care Med. 2010 Mar;38(3):831-7. doi: 10.1097/CCM.0b013e3181cc4a67. PMID 20068467
- [Background] Liao TK, Ho CH, Lin YJ, Cheng LC, Huang HY. Shock index to predict outcomes in patients with trauma following traffic collisions: a retrospective cohort study. Eur J Trauma Emerg Surg. 2024 Oct;50(5):2191-2198. doi: 10.1007/s00068-024-02545-4. Epub 2024 May 31. PMID 38819683
- [Background] Bouzat P, Ageron FX, Brun J, Levrat A, Berthet M, Rancurel E, Thouret JM, Thony F, Arvieux C, Payen JF; TRENAU group. A regional trauma system to optimize the pre-hospital triage of trauma patients. Crit Care. 2015 Mar 18;19(1):111. doi: 10.1186/s13054-015-0835-7. PMID 25887150
- [Background] Baker SP, O'Neill B, Haddon W Jr, Long WB. The injury severity score: a method for describing patients with multiple injuries and evaluating emergency care. J Trauma. 1974 Mar;14(3):187-96. No abstract available. PMID 4814394
- [Background] Rating the severity of tissue damage. I. The abbreviated scale. JAMA. 1971 Jan 11;215(2):277-80. doi: 10.1001/jama.1971.03180150059012. No abstract available. PMID 5107365
- See also: Insee. Statistiques sur les accidents En France. — https://www.insee.fr/fr/statistiques
- See also: Santé publique France. "Traumatismes non intentionnels." Bulletin épidémiologique hebdomadaire. 2023 — https://www.santepubliquefrance.fr
- See also: Trauma center Association of America. Best Practices in Trauma Care — https://www.traumacenters.org
- See also: Santé publique France. "Traumatismes et accidents de la vie courante." Publié le 6 mai 2022 — https://www.santepubliquefrance.fr/maladies-et-traumatismes/traumatismes
- See also: Thèse de Doctorat Université de Rennes 1 — https://dumas.ccsd.cnrs.fr/dumas-00631527
- See also: Thèse de Doctorat en santé Publique - Epidémiologie. Université Paris-Saclay — https://theses.hal.science/tel-03084258
- See also: Thèse de Doctorat Université de Grenoble — https://dumas.ccsd.cnrs.fr/dumas-01119343